CLINICAL TRIAL: NCT01010165
Title: Caractérisation de Nouveaux Biomarqueurs de l'Arthrite Septique Par Technique SELDI-TOF
Brief Title: Determination of New Biomarkers of Septic Arthritis by Surface-Enhanced Laser Desorption/Ionization Time-Of-Flight (SELDI-TOF)
Acronym: NOUBASST
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 0916; 2009-A00810-57 (Registry Identifier: RCB)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2011-12

CONDITIONS: Acute Arthritis
Keywords: acute arthritis; bacteria; crystal arthritis; proteomic; SELDI-TOF
MeSH Terms: conditions — Crystal Arthropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — joint fluid proteom
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- septic arthritis
- crystal arthritis
- rheumatismal disease

SUMMARY:
Septic arthritis is a frequent, potentially disabling and/or life-threatening disease. To diagnose a septic arthritis is a complex procedure, first because of numerous differential diagnoses (such as crystal arthritis), second because of poor sensitivity of initial gram staining (for example after untimely antibiotic therapy).

This protocol will use SELDI-TOF as a tool to analyse joint fluid of patients with various acute, polymorphonuclear-rich arthritis, as to determine specific and sensitive new biomarkers of a septic origin.

Such biomarkers will allow rapid diagnosis of septic arthritis in the first hours of admission.

ELIGIBILITY:
Inclusion Criteria:

* acute arthritis (onset not more than 7 days ago)
* joint fluid leukocyte count : more than 2000/mm3, more than 50% polymorphonuclear

Exclusion Criteria:

* none (apart from unability to accept inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from the Grenoble University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: olivier epaulard, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France